CLINICAL TRIAL: NCT06818279
Title: Compare the Efficacy and Safety of Dabigatran and Enoxaparin in Patients With Portal Vein Thrombosis With Cirrhosis: A Randomized Controlled Study
Brief Title: Compare the Efficacy and Safety of Dabigatran and Enoxaparin in Patients With Portal Vein Thrombosis With Cirrhosis
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-72
Record Dates: First submitted 2025-01-27; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Portal Vein Thrombosis; Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Dabigatran; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enoxaparin (Active Comparator): Enoxaparin Treatment would be given with 1 mg /Kg (100IU/Kg) dose s/c twice daily for 6 months.
  Interventions: Drug: Enoxaparin
- Dabigatran (Experimental): Dabigatran 150 mg BD fixed dose to be given for duration of 6 months.
  Interventions: Drug: Dabigatran

INTERVENTIONS:
Drug: Dabigatran — Dabigatran 150 mg BD fixed dose to be given for duration of 6 months.
  Arms: Dabigatran
Drug: Enoxaparin — Enoxaparin . Treatment would be given with 1 mg /Kg (100IU/Kg) dose s/c twice daily for 6 months.
  Arms: Enoxaparin

SUMMARY:
Portal vein thrombosis (PVT) is prevalent among patients with cirrhosis, and its prevalence rises with the severity of liver disease. Numerous studies have indicated that patients developing PVT experience elevated portal pressure and associated complications, such as increased incidence of variceal bleeding, higher rates of failed variceal bleed control, rebleeding, and short-term mortality. Additionally, the development of PVT adversely affects post-transplant outcomes, correlating with increased 30-day mortality among transplant recipients with PVT. Current guidelines lack clarity regarding the optimal choice of anticoagulation therapy for patients with cirrhosis. This study aims to evaluate the efficacy and safety of enoxaparin and dabigatran in achieving complete recanalization of portal vein thrombosis in cirrhotic patients over a 6-month period.

DETAILED DESCRIPTION:
Study population: Cirrhosis with portal vein thrombosis within 6 months of diagnosis of portal vein thrombus Study design - A prospective, randomized, single center open label study Block Randomization, block size - 10 Study site - Department of Hepatology, ILBS, New Delhi from The study will be conducted on the consecutive patients with liver cirrhosis with portal vein thrombosis.

Study period -1 year Monitoring and assessment

* At enrollment:

  1. Complete history and physical examination
  2. Etiology of cirrhosis
  3. Presenting symptoms
  4. Severity of ascites, Jaundice
  5. Pattern and number of prior decompensation
  6. UGIE and variceal status
  7. Complete physical evaluation
  8. Hemogram, Kidney function test, Liver function test, INR
  9. Ultrasound abdomen with spleno-portal axis doppler / CECT upper abdomen
  10. Fibroscan-liver and spleen
  11. 2D-ECHO, ECG
  12. AFP At follow-up (1month, 3 month, 6 month, 9 month 12month)

  <!-- -->

  1. Complete history and physical examination
  2. Pattern and number of decompensation
  3. MELD, CTP, APRI, ALBI Score
  4. Hemogram, Kidney function test, Liver function test, INR
  5. Ultrasound abdomen with spleno-portal axis doppler / CECT upper abdomen

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Cirrhosis with portal vein thrombosis within 6 months of diagnosis/Symptomatic PVT/PVT in potential transplant recipient.

Exclusion Criteria:

1. Contraindications to anticoagulant therapy, such as active bleeding, recent major surgery, or known hypersensitivity to study medications.
2. CTP >10
3. Hepatocellular carcinoma
4. Tumoral PVT
5. Isolated gastric varices with red colour signs
6. Peptic ulcer disease with large ulcers
7. Pregnant or breastfeeding women
8. Thrombocytopenia (platelet count <50,000/μL)
9. Patients with concurrent acute kidney injury or chronic kidney disease stage 4 or 5
10. Those not giving consent for therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achiving recanalization of Portal Vein Thrombosis (PVT) in cirrhosis patients at 6-months in both groups. | 6 months

SECONDARY OUTCOMES:
Rate of complete recanalization of Portal Vein Thrombosis in cirrhosis patients at 6-months in between groups. | 6 months
Rate of partial recanalization of Portal Vein Thrombosis in cirrhosis patients at 6-months in between groups. | 6 months
Rate of complete recanalization of Portal Vein Thrombosis in cirrhosis patients at 3-months in between groups. | 3 months
Rate of recurrence of Portal Vein Thrombosis at 12 months. | 12 months
Adverse events in both the groups till 6-months | 6 months
Change in CTP scores in both the groups over 12-months | 12-months
Change in MELD scores in both the groups over 12-months | 12-months
Variceal and non-variceal bleeding rates at 6-months and 12-months | 6-months and 12-months
Number of patients with worsening of decompensation events and new onset decompensation events in the two study groups till 12-months | 12-months
  Decompensation events includes any of the one ascites,HE,bleed and jaundice
Baseline parameters for predicting recanalisation of Portal Vein Thrombosis (PVT) at 6 months in both the groups. | 12 months
Baseline parameters for predicting rethrombosis of PVT at 12 months in both the groups. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided